CLINICAL TRIAL: NCT05405088
Title: Identification of Predictive Factors of Postoperative Pain After Oral Surgery From Phenotypic Parameters Easily Accessible Preoperatively
Brief Title: Identification of Predictive Factors of Postoperative Pain After Oral Surgery From Phenotypic Parameters Easily Accessible Preoperatively (PHEDOPO)
Acronym: PHEDOPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RBHP 2021 DEVOIZE 2; 2021-A02885-36 (Other: ANSM)
Record Dates: First submitted 2022-04-05; First posted 2022-06-06 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Pain, Postoperative; Anxiety, Dental
Keywords: Pain; Oral surgery; Postoperative; Gender; Eye color; Blood group; Hair color
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Pain; Coitus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: This is a collection of data from postoperative questionnaires and simple, non-invasive clinical observations. The oral surgery acts in question are performed in daily practice without any change in patient management. The intraoperative data collected come from routine care. Postoperative data (pain and analgesic intake) are collected by self-questionnaires and no visit on purpose is required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label cohort, with short follow-up (Other): This is a collection of data from postoperative questionnaires and simple, non-invasive clinical observations. The oral surgery acts in question are performed in daily practice without any change in patient management. The intraoperative data collected come from routine care. Postoperative data (pain and analgesic intake) are collected by self-questionnaires and no visit on purpose is required.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Pain Sensitive Questionnaire (PSQ) Corah's Dental Anxiety Scale (CDAS) Pain Catastrophizing Scale (PCS) Gender Eye color Hair color Blood group

SUMMARY:
This project aims to study various predictive factors of postoperative pain after oral surgery among different parameters accessible preoperatively, in order to build a predictive model. It also aims to validate the external consistency of the Pain Sensitivity Questionnaire in an odontological context.

DETAILED DESCRIPTION:
This project aims to study various predictive factors of postoperative pain after oral surgery among different phenotypic parameters accessible to preoperative interrogation (anxiety about dental care, personal perception of pain sensitivity, gender, eye color, hair color, blood group) in order to build a predictive model. It also aims to validate the external consistency of the Pain Sensitivity Questionnaire (PSQ) in an odontological context, by studying the relationship between the personal perception of pain sensitivity (measured by the PSQ) and anxiety about dental care (measured by the Corah Dental Anxiety Scale), as well as dramatization in the face of pain (measured by the Pain Catastrophizing Scale).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, male or female, eligible for dental extraction under local anesthesia,

  * either a tooth on the arch,
  * either wisdom tooth(s) (2 homolateral wisdom teeth (maxilla + mandibular) or a mandibular wisdom tooth).
* Fluent in speaking and reading French.
* Able to give informed consent to research.
* Affiliation to a Social Security scheme.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Contraindication to paracetamol, NSAIDs, tramadol, or anesthetic agents local.
* Patient uncooperative, unlikely or unable to comply with all procedures of the protocol.
* Chronic use of opiates, in a therapeutic or illicit context.
* Chronic depression on long-term antidepressants.
* Stomatological pathology that may interfere with the conduct of the intervention or modify the results: insufficient mouth opening, pathologies of the temporal mandibular joints ...
* Active medical pathology, or any medical condition judged by the investigator to be incompatible with the study.
* Patient under guardianship, curatorship or safeguard of justice.
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Postoperative pain Day 1 | Information gathering on the morning of day 1
  The pain will be measured from the collection of an intensity measured on a simple 11-point numerical scale (ENS) ranging from "0 = no pain" to "10 = the worst pain imaginable"
Postoperative pain Day 1 | Information gathering on the evening of day 1
  The pain will be measured from the collection of an intensity measured on a simple 11-point numerical scale (ENS) ranging from "0 = no pain" to "10 = the worst pain imaginable"
Postoperative pain Day 2 | Information gathering on the morning of day 2
  The pain will be measured from the collection of an intensity measured on a simple 11-point numerical scale (ENS) ranging from "0 = no pain" to "10 = the worst pain imaginable"
Postoperative pain Day 2 | Information gathering on the evening of day 2
  The pain will be measured from the collection of an intensity measured on a simple 11-point numerical scale (ENS) ranging from "0 = no pain" to "10 = the worst pain imaginable"
Postoperative pain Day 3 | Information gathering on the morning of day 3
  The pain will be measured from the collection of an intensity measured on a simple 11-point numerical scale (ENS) ranging from "0 = no pain" to "10 = the worst pain imaginable"
Postoperative pain Day 3 | Information gathering on the evening of day 3
  The pain will be measured from the collection of an intensity measured on a simple 11-point numerical scale (ENS) ranging from "0 = no pain" to "10 = the worst pain imaginable"
Postoperative pain Day 4 | Information gathering on the morning of day 4
  The pain will be measured from the collection of an intensity measured on a simple 11-point numerical scale (ENS) ranging from "0 = no pain" to "10 = the worst pain imaginable"
Postoperative pain Day 4 | Information gathering on the evening of day 4
  The pain will be measured from the collection of an intensity measured on a simple 11-point numerical scale (ENS) ranging from "0 = no pain" to "10 = the worst pain imaginable"
Postoperative pain Day 5 | Information gathering on the morning of day 5
  The pain will be measured from the collection of an intensity measured on a simple 11-point numerical scale (ENS) ranging from "0 = no pain" to "10 = the worst pain imaginable"
Postoperative pain Day 5 | Information gathering on the evening of day 5
  The pain will be measured from the collection of an intensity measured on a simple 11-point numerical scale (ENS) ranging from "0 = no pain" to "10 = the worst pain imaginable"

SECONDARY OUTCOMES:
Explanatory variable 1: Pain Sensitive Questionnaire | 1 time only before surgery
  The Pain Sensitivity Questionnaire (PSQ) is a self-administered questionnaire comprising 17 items, each rated from 0 to 10. items n° 3-6-7-10-11-12-14 evoke moderately painful situations (and their sum makes it possible to calculate a "minor" PSQ score), and items n° 1-2-4-8- 15-16-17 evoke clearly painful situations (and their sum makes it possible to calculate a "moderate" PSQ score). The sum of these two scores is the "total" PSQ score. As each response to each item ranges from 0 to 10, the minimum value for all scores is 0, and the maximal ones for the minor, the moderate and the total PSQ scores are respectively 7, 7 and 14. The higher the scores, the higher the sensitivity to pain.
Explanatory variable 2: Corah's Dental Anxiety Scale (CDAS) | 1 time only before surgery
  Corah's Dental Anxiety Scale is based on 4 main questions and calculates a score from 5 to 20 (0-8: no anxiety; 9-12: moderate anxiety; 13-14: high anxiety; 15-20: severe anxiety)
Explanatory variable 3: Pain Catastrophizing Scale (PCS) | 1 time only before surgery
  Pain Catastrophizing Scale is based on 13 questions that cover 3 representative domains of dramatization: exaggeration of the pain felt (magnification), the tendency to constantly meditate on the pain (rumination) and the feeling of abandonment or lack of associated support (helplessness). As each response to each of the 13 responses items ranges from 0 to 4, the minimum value for the PCS score is 0, and the maximal is 52. The higher the score, the higher the level of pain catastrophizing.
Explanatory variable 4: Gender | 1 time only before surgery
  Gender will be determined between male or female subject
Explanatory variable 5: Eye color | 1 time only before surgery
  The color of the iris will be determined by the scale of Martine and Schultz:
  Light tones:
  1-2: Blue 3: Blue gray 4: Gray 5: Blue-gray with yellow/brown spots 6: Grey-green with yellow/brown spots 7: Green 8: Green with yellow/brown spots 9-10-11: Light brown or hazelnut brown
  Dark tones:
  12-13: Brown 14-15: Dark brown to black
Explanatory variable 6: Hair color | 1 time only before surgery
  Hair color will be determined by color:
  Black Brown Blond Red
Explanatory variable 7: Blood group | 1 time only before surgery
  The blood group will be determined by the groups:
  O HAS B AB as well as Rhesus + or -

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Devoize, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France